CLINICAL TRIAL: NCT05692271
Title: Testing a Novel Therapeutic Strategy for Comorbid Post-Traumatic Stress Disorder and Alcohol Use Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 061-2021
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Stress Disorders, Post-Traumatic; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol (Experimental): Medication treatment regimen will consist of 12 weeks of 40 mg immediate-release propranolol BID
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): Matching placebo will be administered BID for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — 40 mg teva-propranolol taken twice daily for 12 weeks
  Arms: Propranolol
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This study evaluates the therapeutic tolerability of the use of Cognitive Processing Therapy (CPT) with propranolol in participants with Posttraumatic Stress Disorder (PTSD) and Alcohol Use Disorder (AUD). The investigators are planning to perform an initial proof -of- concept randomized, placebo- controlled trial evaluating propranolol in participants with PTSD and AUD starting CPT for 12 weeks with three post-treatment follow ups at week-16, week-20, and week-24.

Participants with current diagnosis of PTSD and AUD seeking treatment will be randomized to either a propranolol group (n=24) or placebo group (n=24) after enrollment. All participants will receive CPT for 12 weeks after randomization. Primary outcomes will be measured in both groups at the end of the study (week 12).

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 and 70 years old inclusively
2. Diagnosed with AUD in the past year (according to the Structured Clinical Interview for DSM-5 (SCID)25). This will include active drinkers and recently abstained drinkers.
3. has a minimum of two episodes of heavy drinking (≥5 drinks in a single day for men and ≥4 drinks in a single day for women) in the past 30 days as used in other trials26
4. Diagnosed with current (past 30 days) PTSD with the Clinician- Administered PTSD Scale for DSM-5 (CAPS-5) on screening27
5. On an antidepressant as treatment of PTSD (to ensure safety and homogeneity as PTSD treatment of study population). Antidepressants are the first-line treatment for PTSD as well major depression which commonly comorbid PTSD. The presence of antidepressants in study recruitment criteria will ensure additional safety if the trauma focused therapy triggered emotional distress which could temporarily activate depressive symptoms. The presence of antidepressants in all study participants will also ensure proper evaluation of the effect of propranolol without any confounders effect.
6. Agrees (if the participant is female and of childbearing potential) to use at least one of the following highly effective methods of contraception, such as hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation or alternatively double barrier method.
7. Agrees not to start any other therapy including self-help group during the trial period. Exception will be made for participants who had already started therapy and have been attending the sessions for at least 6 months.
8. Agrees not to start any anti-craving medications for alcohol use during the trial period. Exception will be made for participants who were already taking an anti-craving medication for at least 6 months.
9. Able to speak and read in English

Exclusion Criteria:

1. Diagnosed with a severe or unstable medical illness that precludes safe participation in the study as per study physician, including contraindications to propranolol administration such as asthma, diabetes, arrhythmia or congestive heart failure
2. Diagnosed with psychotic disorder or bipolar disorder
3. The use of alcohol abstinence medications within the past month
4. Current moderate or severe substance use disorder (excluding alcohol, cannabis, tobacco and caffeine)
5. A basal systolic blood pressure < 100 mm Hg or basal heart rate < 55 beats/minute
6. Pregnant or breastfeeding women
7. Individuals with known hypersensitivity to propranolol
8. Individuals with current use of medication that might interact adversely with propranolol such as anti-arrhythmic medication or calcium channel blockers
9. Current suicidality risk as indicated during the conduct of the Columbia Suicide Severity Rating Scale (C-SSRS) with concurrence after a study physician's evaluation if the response to C-SSRS questions 1 or 2 is "yes"28
10. Any participant known to have non-allergic bronchospasm such as chronic bronchitis, emphysema, bronchiectasis, hypotension, metabolic acidosis, severe peripheral arterial circulatory disturbance, untreated phaeochromocytoma, Prinzmetal's angina
11. Any participant with known hypersensitivity to any ingredient in the formulation, including any non-medicinal ingredient, or component of the container.
12. Any participant using catecholamine depletion drugs such as reserpine or guanethidine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Number of CPT sessions attended | 12 weeks
  Number of CPT (therapy) sessions attended by participants

SECONDARY OUTCOMES:
CAPS-5 total symptom severity score | 12 weeks
  PTSD symptoms measured using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) scores at baseline, midpoint (week-6) and endpoint (week 12); the CAPS-5 total symptom severity score is the sum of severity (rated 0-4) on 20 individual items, where a higher score indicates greater symptom severity
Number of drinks per week (TLFB) | 12 weeks
  Alcohol consumption to be monitored using the timeline follow-back (TLFB)
Percent heavy drinking days (TLFB) | 12 weeks
  Percent heavy drinking days will be measured weekly. A "heavy drinking day" will be defined as 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
Alcohol craving | 12 weeks
  Alcohol craving will be assessed using the Penn Alcohol Craving Scale (PACS), which includes five items scored on a Likert scale from 0 to 6 Min score=0, max score=30, higher scores indicate greater craving

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hassan, MD, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided